CLINICAL TRIAL: NCT02848638
Title: Pair Production PET Imaging to Detect Particle Distribution in Patients Undergoing Yttrium-90 Radioembolization With Large Hepatocellular Carcinomas or Associated Portal Vein Thrombosis
Brief Title: Pair Production PET Imaging to Detect Particle Distribution in Patients Undergoing Yttrium-90 Radioembolization
Acronym: PET-Y90
Status: Completed | Type: Observational
Sponsor: University of Washington (Other)
Responsible Party: Principal Investigator, Siddharth A. Padia, Associate Professor, University of Washington
Other Study IDs: 42413
Record Dates: First submitted 2016-07-26; First posted 2016-07-28 (Estimated); Last update posted 2018-08-02 (Actual); Status verified 2018-07

CONDITIONS: Carcinoma, Hepatocellular
Keywords: PET, Yttrium-90
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The primary goal of the study is to see if the PET/CT will be able to determine the precise location of the Y-90 particles within the liver and within the tumors. We hope to use this information in order to see if these particles distribute evenly throughout large tumors or if the particles go into the tumor which is located in the portal vein.

The secondary goals are threefold. First correlate the distribution of Y90 particles (as demonstrated by PET/CT) with the degree of dead-tumor tissue. Second, see if there is a difference in the Y90 particle's distribution when a low particle load (1-3 million particles) is used compared to when a high particle load (6-8 million particles) is used. Lastly, compare the sensitivity of standard imaging ( bremsstrahlung imaging) currently being used for the Yttrium-90 angioembolization procedure to the sensitivity of the pair production PET research imaging.

ELIGIBILITY:
Inclusion Criteria:

1. UWMC patients over 18 years of age
2. Presence of hepatocellular carcinoma greater than 5 cm OR presence of tumor-associated portal vein thrombosis.
3. Currently undergoing treatment with Yttrium-90 Radioembolization
4. Able to sign informed consent

Exclusion Criteria:

1. Patients who are not undergoing treatment with Yttrium-90 Radioembolization
2. Patients unable to provide informed consent

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients (18-85 years old), who have hepatocellular carcinoma with tumors that are greater than 5 cm or have tumor-associated portal vein thrombosis. The patients are currently undergoing treatment with Yttrium-90 Radioembolization, as part of their clinical care.
Sampling Method: Non-Probability Sample
Enrollment: 35 (Actual)
Dates: Start 2012-07 (Actual); Primary Completion 2016-03 (Actual); Study Completion 2018-03-31 (Actual)

PRIMARY OUTCOMES:
Degree and distribution of Y90 particle uptake | Within one year of Enrollment completion
  To use pair production PET/CT in order to determine the degree and distribution of Y90 particle uptake in patients with large (>5cm) liver tumors or patients with tumor-associated portal vein thrombosis.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Chan KT, Alessio AM, Johnson GE, Vaidya S, Kwan SW, Monsky W, Wilson AE, Lewis DH, Padia SA. Hepatotoxic Dose Thresholds by Positron-Emission Tomography After Yttrium-90 Radioembolization of Liver Tumors: A Prospective Single-Arm Observational Study. Cardiovasc Intervent Radiol. 2018 Sep;41(9):1363-1372. doi: 10.1007/s00270-018-1949-5. Epub 2018 Apr 12. PMID 29651580